CLINICAL TRIAL: NCT06711406
Title: The Effect of Attention on Postural Control
Status: Completed | Type: Observational
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Çiğdem Yazıcı Mutlu, assistant prof, Yeditepe University
Other Study IDs: Effect of Attention on Posture
Record Dates: First submitted 2024-11-25; First posted 2024-12-02 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: ADHD - Attention Deficit Disorder with Hyperactivity; Postural Instability
Keywords: ADHD; Posture; Attention; Balance; Dual task
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ASRS-5 score above 14: This group consists of participants who have a score of 14 and above on the Adult ADHD Self-Report Scale (ASRS-5). Participants with these scores are more susceptible to ADHD. The group does two cognitive tests, the Sustained Attention to Response Test (SART) TEST. Furthermore, the assessment of their Postural Control is conducted using a force plate.
- ASRS-5 score Below 14: This group consists of participants who have a score below 14 on the Adult ADHD Self-Report Scale (ASRS-5). Participants with these scores are less susceptible to ADHD. Participants with these scores are more vulnerable to ADHD. The group does two cognitive tests, the Sustained Attention to Response Test (SART) TEST. Furthermore, the assessment of their Postural Control is conducted using a force plate.

SUMMARY:
Objective: This study investigates the relationship between postural control and sustained attention in individuals with probable ADHD. Motor control issues, including balance deficits, are observed in 30-50% of children with ADHD. These deficits may extend into adulthood, yet research on postural control in adults with ADHD is limited. This study aims to address this gap by exploring the connection between attention and postural stability in adults with ADHD.

Background: ADHD is a neurodevelopmental disorder characterized by inattention, hyperactivity, and impulsivity, affecting both children and adults. Studies have shown that postural control relies on coordinated functioning of sensory and neuromotor systems, which ADHD may impact. In children, postural challenges are more pronounced in conditions requiring complex sensory integration. However, research on adults with ADHD is sparse, though preliminary findings suggest postural instability and possible links to cerebellar differences.

Methodology: The study evaluates sustained attention and postural control in adults with ADHD, using the Adult ADHD Screening Scale (ASRS-5) and postural stability assessments under dual-task conditions. By examining attention-driven postural responses, the study contributes to developing therapeutic balance protocols for individuals with ADHD.

Hypotheses:

H0: No relationship exists between postural control and sustained attention in individuals with ADHD.

H1: A relationship exists between postural control and sustained attention in individuals with ADHD.

Significance: This study contributes to a better understanding of the neurophysiological links

ELIGIBILITY:
Inclusion Criteria:

* Volunteers between 18-30-year-olds
* Not having any problems with balance

Exclusion Criteria:

* Having a physical injury in the last 6 months (such as ankle sprain)
* Having any neurological disorder
* Exercising regularly for the last 12 months

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study was planned with healthy young volunteers (18-30-year-olds) who have the potential to have ADHD. Our target population was university students.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Postural Control: Prokin PK 252. | 30 minutes
  The Prokin device (Prokin PK 252) is a proprioceptive system for static and dynamic balance assessment and training. The device shows multiple programs for balance assessment and treatment. For this experiment, the "Static Stability Assessment Program" will be chosen to provide detailed and precise data of each participant while static standing through the stabilometry platform and the sensor placed on the trunk. Stabilometry allows participants to be evaluated by detecting the oscillation of the Centre of Pressure (CoP) during static standing. The platform of the Prokin device will calculate the CoP sways of the participants and the postural control data will be transferred to the computer screen. The assessment will be done in two conditions: a two-foot standing position without stimulus (eyes open, eyes closed), and a two-foot standing position with dual-task (eyes open, eyes closed). The dual-task procedure involves instructing participants to count down from 100 by 3.

SECONDARY OUTCOMES:
Cognitive tests: Sustained Attention to Response Task (SART): | 5 minutes
  The Sustained Attention to Response Task (SART) is a computer-based task where participants need to refrain from responding to a rare target (the digit 3) embedded within a series of more frequent non-targets (0-2, 4-9). Participants were instructed to prioritize both accuracy and speed in completing the task.

CONTACTS AND LOCATIONS:
Overall Officials: Çiğdem Yazıcı Mutlu, PhD, Study Director — Yeditepe University
Locations (1):
- Yeditepe University, Istanbul, Ataşehit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided